CLINICAL TRIAL: NCT01511263
Title: A Phase II Open-label Randomized Study of Dietary Supplement With Epigallocatechin Gallate (EGCG) to Improve Cardiac Dysfunction in Patients With AL Amyloidosis Who do Not Require Chemotherapy (EpiCardiAL)
Brief Title: Epigallocatechingallate (EGCG) in Cardiac AL Amyloidosis
Acronym: EpiCardiAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giampaolo Merlini, Director, Amyloidosis Research and Treatment Center, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-006-IT
Record Dates: First submitted 2012-01-10; First posted 2012-01-18 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Primary Amyloidosis of Light Chain Type
Keywords: Epigallocatechin gallate; AL amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): The patients will be divided into 4 strata according to cardiac dysfunction and to the quality of hematologic response. After stratification the patients will be randomized (1:1) within each stratum to receive Standard Therapy alone (Arm A) or Standard Therapy plus Investigational Drug (Arm B).
  Interventions: Drug: Diuretics (plus antiarrhythmic drugs, i.e. amiodarone, in case of complex ventricular arrhithmias)
- Arm B (Experimental): The patients will be divided into 4 strata according to cardiac dysfunction and to the quality of hematologic response. After stratification the patients will be randomized (1:1) within each stratum to receive Standard Therapy alone (Arm A) or Standard Therapy plus Investigational Drug (Arm B)
  Interventions: Drug: Diuretics (plus antiarrhythmic drugs, i.e. amiodarone, in case of complex ventricular arrhythmias) plus EGCG

INTERVENTIONS:
Drug: Diuretics (plus antiarrhythmic drugs, i.e. amiodarone, in case of complex ventricular arrhithmias) — Antiarrhythmic drugs (i.e. amiodarone), angiotensins which transform inhibitor enzymes, and/or beta-blockers if tolerated.
  Arms: Arm A
Drug: Diuretics (plus antiarrhythmic drugs, i.e. amiodarone, in case of complex ventricular arrhythmias) plus EGCG — Antiarrhythmic drugs (i.e. amiodarone), angiotensins which transform inhibitor enzymes, and/or beta-blockers if tolerated.
  EGCG, 675 mg/day, oral, for one year.
  Arms: Arm B

SUMMARY:
In a proportion of patients with AL amyloidosis there is no improvement of cardiac function despite hematologic response to treatment. The aim of the study is to assess whether treatment with EGCG increases the rate of cardiac response in patients with AL amyloidosis who completed chemotherapy.

DETAILED DESCRIPTION:
This will be a phase II open-label randomized trial. Patients with AL amyloidosis and cardiac involvement who have achieved at least partial hematologic response after chemotherapy will be randomized to receive standard supportive therapy (SST) or SST plus Epigallocatechin gallate (EGCG). After giving written informed consent, the patients will be evaluated for eligibility. Briefly, the subjects with a biopsy-proven diagnosis of AL amyloidosis who achieved at least partial response after chemotherapy, who are not planned to receive further chemotherapy and who have significant cardiac dysfunction will be considered eligible. The patients will be stratified according to the quality of hematologic response and to the severity of cardiac involvement. Following stratification, the patients will be randomized to receive SST or SST plus EGCG. The study comprises 3 periods: screening (including stratification and randomization), treatment (with evaluations of response every 2 months) followed by the end-of-treatment evaluation and follow-up. Therapy will continue for up to 1 year. After treatment patients will be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AL amyloidosis.
* Age ≥18 years.
* The patients must have been treated for AL amyloidosis attaining hematologic response.
* Evidence of cardiac involvement at echocardiography (mean left ventricular wall thickness >12 mm in the absence of other causes).
* NT-proBNP ≥650 ng/L

Exclusion Criteria:

* Non-AL (e.g. familial, senile) amyloidosis.
* Concomitant non-amyloid related clinically significant cardiac diseases.
* Need of further chemotherapy for AL amyloidosis.
* Estimated glomerular filtration rate (eGFR) <30 mL/min per 1.73 m2.
* Uncontrolled infection.
* Inability to give informed consent.
* Previous or ongoing psychiatric illness (excluding reactive depression).
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cardiac response | 6 months
  The primary objective is to assess whether treatment with EGCG increases the rate of cardiac response following chemotherapy in patients with AL amyloidosis. The primary endpoint is cardiac response at 6 months.

SECONDARY OUTCOMES:
Rate of adverse events | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.
Rate of cardiac progression | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.
Time to cardiac progression | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.
Rate of cardiac events | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.
Time to cardiac events | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.
Survival | 6 months
  The secondary objectives are to assess the safety of EGCG in cardiac AL amyloidosis, to determine whether EGCG can prevent or delay cardiac progression and to compare survival of patients receiving EGCG compared to subjects receiving SST.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico S.Matteo, Pavia, Italy

REFERENCES:
- [Background] Dispenzieri A, Gertz MA, Kyle RA, Lacy MQ, Burritt MF, Therneau TM, Greipp PR, Witzig TE, Lust JA, Rajkumar SV, Fonseca R, Zeldenrust SR, McGregor CG, Jaffe AS. Serum cardiac troponins and N-terminal pro-brain natriuretic peptide: a staging system for primary systemic amyloidosis. J Clin Oncol. 2004 Sep 15;22(18):3751-7. doi: 10.1200/JCO.2004.03.029. PMID 15365071
- [Background] Hunstein W. Epigallocathechin-3-gallate in AL amyloidosis: a new therapeutic option? Blood. 2007 Sep 15;110(6):2216. doi: 10.1182/blood-2007-05-089243. No abstract available. PMID 17785589
- [Background] Mereles D, Buss SJ, Hardt SE, Hunstein W, Katus HA. Effects of the main green tea polyphenol epigallocatechin-3-gallate on cardiac involvement in patients with AL amyloidosis. Clin Res Cardiol. 2010 Aug;99(8):483-90. doi: 10.1007/s00392-010-0142-x. Epub 2010 Mar 10. PMID 20221615
- [Background] Mereles D, Wanker EE, Katus HA. Therapy effects of green tea in a patient with systemic light-chain amyloidosis. Clin Res Cardiol. 2008 May;97(5):341-4. doi: 10.1007/s00392-008-0649-6. Epub 2008 Mar 3. No abstract available. PMID 18317666
- [Background] Merlini G, Palladini G. Amyloidosis: is a cure possible? Ann Oncol. 2008 Jun;19 Suppl 4:iv63-6. doi: 10.1093/annonc/mdn200. No abstract available. PMID 18519408
- [Background] Palladini G, Barassi A, Klersy C, Pacciolla R, Milani P, Sarais G, Perlini S, Albertini R, Russo P, Foli A, Bragotti LZ, Obici L, Moratti R, Melzi d'Eril GV, Merlini G. The combination of high-sensitivity cardiac troponin T (hs-cTnT) at presentation and changes in N-terminal natriuretic peptide type B (NT-proBNP) after chemotherapy best predicts survival in AL amyloidosis. Blood. 2010 Nov 4;116(18):3426-30. doi: 10.1182/blood-2010-05-286567. Epub 2010 Jul 19. PMID 20644111
- [Background] Palladini G, Campana C, Klersy C, Balduini A, Vadacca G, Perfetti V, Perlini S, Obici L, Ascari E, d'Eril GM, Moratti R, Merlini G. Serum N-terminal pro-brain natriuretic peptide is a sensitive marker of myocardial dysfunction in AL amyloidosis. Circulation. 2003 May 20;107(19):2440-5. doi: 10.1161/01.CIR.0000068314.02595.B2. Epub 2003 Apr 28. PMID 12719281
- See also: Related Info — http://www.amiloidosi.it/